CLINICAL TRIAL: NCT04891705
Title: Point of Care Ultrasound Lung Artificial Intelligence (AI) Validation Data Collection Study
Acronym: AI
Status: Completed | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Other Study IDs: US-Lung AI-11237
Record Dates: First submitted 2021-05-13; First posted 2021-05-18 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-11

CONDITIONS: Pleural Effusion; Lung Consolidation
Keywords: Artificial Intelligence; Diagnostics
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Pleural Effusion: Adult and pediatric subjects with suspicion of pleural effusion
  Interventions: Device: Lung Ultrasound Scan
- Lung Consolidation: Adult and pediatric subjects with suspicion of lung consolidation
  Interventions: Device: Lung Ultrasound Scan

INTERVENTIONS:
Device: Lung Ultrasound Scan — Ultrasound scan of subjects in up to 14 lung zones

SUMMARY:
This study is being conducted to collect image data and relevant clinical data from medical records of patients with suspicion of lung consolidation or pleural effusion. The information will be used to test the performance of Artificial Intelligence (AI) in identification of features associated with the above lung conditions.

DETAILED DESCRIPTION:
This is a prospective, observational, multi-center, post-market clinical study. Enrollment will continue (up to a maximum of 500 adult subjects and up to 300 pediatric subjects) until diagnostic LUS exams are acquired for each of the following groups:

Approximately 500 Adult subjects targeting:

* Approximately 175 exams from patients positive for lung consolidation
* Approximately 175 exams from patients positive for pleural effusion
* Approximately 150 exams from patients negative for both conditions

Approximately 300 pediatric subjects targeting:

* Approximately 150 exams from patients positive for lung consolidation
* Approximately 150 exams from patients negative for lung consolidation

ELIGIBILITY:
Inclusion Criteria:

1. Subjects presenting to the Emergency Department, admitted to the hospital, or seen in the outpatient setting with suspicion of pleural effusion or lung consolidation who received chest imaging to include chest X-ray or CT, or for whom chest X-ray or CT are planned.

   Suspicion of pleural effusion or lung consolidation may be based upon imaging findings or presentation of symptoms including (but not limited to) dyspnea, hypoxia, tachypnea, rales, or dullness.
2. All attempts should be made for subjects to undergo scanning of 14 lung zones (adults) and 12 lung zones (pediatrics). Attempts should also be made to capture all required lung zones in adults and pediatrics. Instances where all zones cannot be captured need to be documented and reason for inability to scan them provided in EDC. See Section 8.1.3 Lung Ultrasound Exams.
3. Subject is willing to provide informed consent (or assent where age appropriate) to participate in the study. Subjects under 18 years of age require informed consent of a parent or guardian and assent as required by institutional IRB.
4. Weight of subject is greater than or equal to 10 kg.

Exclusion Criteria:

1. Subject has pathology precluding safe and pain-free ultrasound probe placement such as burn, significant soft tissue injury or surgical incisions.
2. Current imprisonment.
3. Pregnancy (self-reported)
4. Subjects with breast implants
5. Prior pleurodesis procedure.
6. History of severe lung disease and home oxygen use
7. Presence of subcutaneous air that precludes imaging
8. Body Mass Index (BMI) > 40
9. Significant scoliosis (Cobb angle ≥ 20 degrees).
10. Pediatric subjects with chronic lung diseases other than asthma.
11. Pediatric subjects on chronic respiratory support (i.e., nasal canula, CPAP, BiPAP, or tracheostomy).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult subjects with suspicion of pleural effusion or lung consolidation will be enrolled in the study. In addition, pediatric subjects with suspicion of lung consolidation (with weight of at least 10 kg) will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 554 (Actual)
Dates: Start 2021-09-11 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
The study data will be used to support future performance assessments for Artificial Intelligence based algorithms as described by FDA guidance for Computer Assisted Detection and Diagnostic Devices | Discharge up to 30 days (Single visit)

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Kruecker, Study Director — Philips Healthcare
Locations (5):
- United States (5):
  - Arizona Emergency Medical Research Center, Tucson, Arizona
  - University of Colorado Hospital, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina